CLINICAL TRIAL: NCT06226194
Title: Genetic Susceptibility to Predict Weight Loss After Bariatric Surgery
Acronym: GENBASU
Status: Recruiting | Type: Observational
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Collaborators: ISCIII (Unknown)
Responsible Party: Principal Investigator, Albert Lecube Torello, Head of Endocrinology Department Arnau de Vilanova University Hospital, Institut de Recerca Biomèdica de Lleida
Other Study IDs: IRBLleida
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid; Genetic Predisposition; Metabolic Syndrome; Weight Loss
MeSH Terms: conditions — Obesity, Morbid; Genetic Predisposition to Disease; Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Saliva and peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Lleida: Saliva sample collection and questionnaire
- Barcelona: Saliva sample collection and questionnaire
- Madrid: Saliva sample collection and questionnaire
- Málaga: Saliva sample collection and questionnaire
- Santiago de Compostela: Saliva sample collection and questionnaire
- Pamplona: Saliva sample collection and questionnaire
- León: Saliva sample collection and questionnaire
- A Coruña: Saliva sample collection and questionnaire
- Mallorca: Saliva sample collection and questionnaire
- Tenerife: Saliva sample collection and questionnaire
- Las Palmas: Saliva sample collection and questionnaire

SUMMARY:
Obesity is a complex chronic disease, in which both genetic and environmental factors are involved, that shows a great heterogeneity in the response to different weight loss programs. Identifying patients as responder or no responder to the different obesity treatment options is a concept of great interest, both due to the high prevalence of obesity and its high consumption of resources. More than 500,000 surgeries are performed every year around the world, of which approximately 30% will present unsatisfactory results.

The general objective is to carry out a multi-omics approach for the discovery and validation of markers of weight response to bariatric surgery (BS) in a large sample of people with severe obesity (n=6,966 men and women who underwent sleeve gastrectomy or gastric bypass, including an additional external validation set). Thus, the investigators want to know the integrated contribution of several genomic markers (Genome Wide Association study, GWAs), new clinical and analytical variables (human exposome concept) and gender perspective to the prediction of response to the intervention at 12 month and its long-term longitudinal maintenance (3 years). The investigators intend, therefore, to provide new evidence to advance towards precision medicine. The investigators will focus our attention also on identifying those patients who, after being classified at the weight loss nadir as responders experienced weight regain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 65 at the time of surgery
* SG or RYBP as bariatric procedure.
* With a BMI≥35.0 kg/m2 with one or more comorbidities or a BMI>40.0 kg/m2 at the time of surgery.
* Provision of an informed consent form signed and personally dated by the patient.
* With available baseline data (anthropometric, analytical, surgical procedure, pharmacological therapies, and obesity-related comorbidities).

Exclusion Criteria:

* Any previous gastrointestinal surgery
* Treatment with any approved antiobesity drug in Spain (orlistat, liraglutide 3.0 mg and/or naltrexone/bupropion extended release) or systemic glucocorticoids for more than 4 consecutive weeks during the 3 years following BS
* End stage kidney disease (eGFR <15 ml/min/1.73m2) or liver cirrhosis at baseline
* Patients who developed any major medical conditions that limits the practice of a healthy life within normal limits (advanced cardiovascular disease or heart failure, stroke with neurological sequelae, chronic pulmonary obstructive disease with dyspnea at minimal exertion, severe joint pathology, end stage renal failure, or active cancer)
* Known type 1 diabetes or LADA diabetes
* Women who become pregnant during the follow-up period
* Current drug or alcohol abuse
* Uncontrolled psychiatric illness or eating disorders developed during the follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter retrospective study will be aimed at 6,966 obese patients undergoing BS, whose surgical technique (sleeve gastrectomy vs gastric bypass) has been performed at least 3 years before, evaluating the best combination of genetic and exposomal characteristics (clinical and analytical) that will predict which patients will be responders and non-responders in terms of weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 6966 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Genomic markers that can predict the weight change response to bariatric surgery | 3 years
  Percentage of initial weight change

SECONDARY OUTCOMES:
Genomic markers that can predict comorbidities response to bariatric surgery | 3 years
  Type 2 diabetes mellitus, sleep apnea, fatty liver

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lecube Torelló, PhD, Study Chair — Institut de Recerca Biomèdica de Lleida; Rafael Simo, PhD, Study Director — Vall d'Hebron Research Institute; Miguel Angel Rubio, PhD, Principal Investigator — Instituto de Investigación Sanitaria Hospital Clínico San Carlos; Francisco Tinahones, PhD, Principal Investigator — Instituto de Investigación Biomédica de Málaga; Javier Escalada, PhD, Principal Investigator — Clínica Universidad de Navarra Institute
Locations (1):
- IRBLleida, Lleida, Leida, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Breton I, de Hollanda A, Vilarrasa N, Rubio Herrera MA, Lecube A, Salvador J, Garcia-Luna PP, Tinahones FJ, Sanchez Santos R, Gomez Huelgas R, Carretero Gomez J, Moize V, Polo Garcia J, Tranche Iparraguirre S, Fernandez-Pro Ledesma A, Escalada J; representing SEEN, SEEDO, SECO, SEMI, SEDYN, SEMERGEN, semFYC and SEMG. Obesity and COVID-19. A necessary position statement. Endocrinol Diabetes Nutr (Engl Ed). 2021 Oct;68(8):573-576. doi: 10.1016/j.endien.2021.02.004. Epub 2021 Nov 18. No abstract available. PMID 34872641
- [Background] Ballesteros Pomar MD, Vilarrasa Garcia N, Rubio Herrera MA, Barahona MJ, Bueno M, Caixas A, Calanas Continente A, Ciudin A, Cordido F, de Hollanda A, Diaz MJ, Flores L, Garcia Luna PP, Garcia Perez-Sevillano F, Goday A, Lecube A, Lopez Gomez JJ, Minambres I, Morales Gorria MJ, Morinigo R, Nicolau J, Pellitero S, Salvador J, Valdes S, Breton Lesmes I. The SEEN comprehensive clinical survey of adult obesity: Executive summary. Endocrinol Diabetes Nutr (Engl Ed). 2021 Feb;68(2):130-136. doi: 10.1016/j.endinu.2020.05.003. Epub 2020 Sep 12. English, Spanish. PMID 32933882
- [Background] Beisani M, Sabench Pereferrer F, Vilallonga R, Gonzalez Lopez O, Molina Lopez A, Del Castillo Dejardin D, Garcia Ruiz de Gordejuela A, Fort Lopez-Barajas JM, Armengol Carrasco M; Members of the Obesity Section of the Spanish Surgical Association Collaborative Group. Seeking an Initial-Weight-Independent Metric in a Mediterranean Cohort of Gastric Bypass Patients: the %AWL Revisited. Obes Surg. 2021 Apr;31(4):1524-1532. doi: 10.1007/s11695-020-05154-3. Epub 2021 Jan 4. PMID 33398625
- [Background] Caixas A, Villaro M, Arraiza C, Montalva JC, Lecube A, Fernandez-Garcia JM, Corio R, Bellido D, Llisterri JL, Tinahones FJ. SEEDO-SEMERGEN consensus document on continuous care of obesity between Primary Care and Specialist Hospital Units 2019. Med Clin (Barc). 2020 Sep 25;155(6):267.e1-267.e11. doi: 10.1016/j.medcli.2019.10.014. Epub 2020 Feb 17. English, Spanish. PMID 32081378
- [Background] Martinez-Ortega AJ, Olveira G, Pereira-Cunill JL, Arraiza-Irigoyen C, Garcia-Almeida JM, Irles Rocamora JA, Molina-Puerta MJ, Molina Soria JB, Rabat-Restrepo JM, Rebollo-Perez MI, Serrano-Aguayo MP, Tenorio-Jimenez C, Vilches-Lopez FJ, Garcia-Luna PP. Recommendations Based on Evidence by the Andalusian Group for Nutrition Reflection and Investigation (GARIN) for the Pre- and Postoperative Management of Patients Undergoing Obesity Surgery. Nutrients. 2020 Jul 6;12(7):2002. doi: 10.3390/nu12072002. PMID 32640531
- [Background] Vilallonga R, Pereira-Cunill JL, Morales-Conde S, Alarcon I, Breton I, Dominguez-Adame E, Ferrer JV, Ruiz-de-Gordejuela AG, Goday A, Lecube A, Garcia-Almenta EM, Rubio MA, Tinahones FJ, Garcia-Luna PP. A Spanish Society joint SECO and SEEDO approach to the Post-operative management of the patients undergoing surgery for obesity. Obes Surg. 2019 Dec;29(12):3842-3853. doi: 10.1007/s11695-019-04043-8. PMID 31342249
- [Background] Lecube A, Monereo S, Rubio MA, Martinez-de-Icaya P, Marti A, Salvador J, Masmiquel L, Goday A, Bellido D, Lurbe E, Garcia-Almeida JM, Tinahones FJ, Garcia-Luna PP, Palacio E, Gargallo M, Breton I, Morales-Conde S, Caixas A, Menendez E, Puig-Domingo M, Casanueva FF. Prevention, diagnosis, and treatment of obesity. 2016 position statement of the Spanish Society for the Study of Obesity. Endocrinol Diabetes Nutr. 2017 Mar;64 Suppl 1:15-22. doi: 10.1016/j.endonu.2016.07.002. Epub 2016 Aug 16. No abstract available. English, Spanish. PMID 27543006
- [Background] Yarnoz-Esquiroz P, Olazaran L, Aguas-Ayesa M, Perdomo CM, Garcia-Goni M, Silva C, Fernandez-Formoso JA, Escalada J, Montecucco F, Portincasa P, Fruhbeck G. 'Obesities': Position statement on a complex disease entity with multifaceted drivers. Eur J Clin Invest. 2022 Jul;52(7):e13811. doi: 10.1111/eci.13811. Epub 2022 May 12. PMID 35514242
- [Background] Linares-Pineda TM, Boughanem H, Gutierrez-Repiso C, Macias-Gonzalez M, Andres-Leon E, Rojo-Martinez G, Valdes S, Tinahones FJ, Morcillo S. Epigenetic changes in the metabolically healthy obese: A case-control versus a prospective study. Eur J Clin Invest. 2022 Aug;52(8):e13783. doi: 10.1111/eci.13783. Epub 2022 Apr 11. No abstract available. PMID 35342930
- [Background] Martinez MC, Meli EF, Candia FP, Filippi F, Vilallonga R, Cordero E, Hernandez I, Eguinoa AZ, Burgos R, Vila A, Simo R, Ciudin A. The Impact of Bariatric Surgery on the Muscle Mass in Patients with Obesity: 2-Year Follow-up. Obes Surg. 2022 Mar;32(3):625-633. doi: 10.1007/s11695-021-05815-x. Epub 2021 Nov 30. PMID 34846686
- [Background] Lecube A, Ciudin A. A long and stony road to the correct treatment of obesity. Med Clin (Barc). 2021 Aug 27;157(4):176-177. doi: 10.1016/j.medcli.2021.06.004. Epub 2021 Jul 10. No abstract available. English, Spanish. PMID 34253348
- [Background] Torrego-Ellacuria M, Barabash A, Larrad-Sainz A, Hernandez-Nunez GM, Matia-Martin P, Perez-Ferre N, Marcuello C, Sanchez-Pernaute A, Torres AJ, Calle-Pascual AL, Rubio MA. Weight Regain Outcomes After Bariatric Surgery in the Long-term Follow-up: Role of Preoperative Factors. Obes Surg. 2021 Sep;31(9):3947-3955. doi: 10.1007/s11695-021-05497-5. Epub 2021 Jun 19. PMID 34146246
- [Background] Gutierrez-Repiso C, Linares-Pineda TM, Gonzalez-Jimenez A, Aguilar-Lineros F, Valdes S, Soriguer F, Rojo-Martinez G, Tinahones FJ, Morcillo S. Epigenetic Biomarkers of Transition from Metabolically Healthy Obesity to Metabolically Unhealthy Obesity Phenotype: A Prospective Study. Int J Mol Sci. 2021 Sep 27;22(19):10417. doi: 10.3390/ijms221910417. PMID 34638758
- [Background] Ciudin A, Fidilio E, Gutierrez-Carrasquilla L, Caixas A, Vilarrasa N, Pellitero S, Simo-Servat A, Vilallonga R, Ruiz A, de la Fuente M, Luna A, Sanchez E, Rigla M, Hernandez C, Salas E, Simo R, Lecube A. A Clinical-Genetic Score for Predicting Weight Loss after Bariatric Surgery: The OBEGEN Study. J Pers Med. 2021 Oct 17;11(10):1040. doi: 10.3390/jpm11101040. PMID 34683180
- [Background] Nicolau J, Dotres K, Ayala L, Rodriguez I, Pascual S, Sanchis P, Bonet A, Tamayo MI, Arteaga M, Fortuny R, Cifuentes A, Masmiquel L. Long-Term Prevalence of Food Addiction Among Bariatric Surgery Patients: Influence on Metabolic and Psychological Outcomes. Metab Syndr Relat Disord. 2021 Apr;19(3):152-158. doi: 10.1089/met.2020.0079. Epub 2021 Feb 18. PMID 33601956
- [Background] Fidilio E, Comas M, Giribes M, Cardenas G, Vilallonga R, Palma F, Pelaez RB, Simo R, Ciudin A. Evaluation of Resting Energy Expenditure in Subjects with Severe Obesity and Its Evolution After Bariatric Surgery. Obes Surg. 2021 Oct;31(10):4347-4355. doi: 10.1007/s11695-021-05578-5. Epub 2021 Aug 3. PMID 34345955
- [Background] Cornejo-Pareja I, Molina-Vega M, Gomez-Perez AM, Damas-Fuentes M, Tinahones FJ. Factors Related to Weight Loss Maintenance in the Medium-Long Term after Bariatric Surgery: A Review. J Clin Med. 2021 Apr 16;10(8):1739. doi: 10.3390/jcm10081739. PMID 33923789
- [Background] Alvarez-Bermudez MD, Martin-Reyes F, Ocana-Wilhelmi L, Moreno-Ruiz FJ, Torres JA, Fernandez-Garcia D, Valdes S, Moreno-Morales N, Garcia-Fuentes E, Tinahones FJ, Garrido-Sanchez L. Variables Associated with Short-Term Weight Loss in a Cohort of Patients with Morbid Obesity According to Age and Three Types of Bariatric Surgery. J Clin Med. 2020 Nov 2;9(11):3537. doi: 10.3390/jcm9113537. PMID 33147793
- [Background] Hollanda A, Lecube A, Rubio MA, Sanchez E, Vilarrasa N, Oliva JG, Fernandez-Soto ML, Salas-Salvado J, Ballesteros-Pomar MD, Ciudin A, Torres F, Vidal C, Morales MJ, Valdes S, Pellitero S, Minambres I, Masmiquel L, Goday A, Suarez L, Flores L, Bueno M, Caixas A, Breton I, Camara R, Olbeyra R, Penso R, Jose de la Cruz M, Simo-Servat A, Pereyra-Garcia FM, Lopez-Mezquita ET, Gils A, Fidilio E, Bandres O, Martinez A, Abuin J, Marques-Pamies M, Tuneu L, Arteaga M, Castaner O, Goni F, Arrizabalaga C, Botana MA, Calanas A, Rebollo A. New Metrics to Assess Type 2 Diabetes After Bariatric Surgery: The "Time-Within-Remission Range". J Clin Med. 2020 Apr 9;9(4):1070. doi: 10.3390/jcm9041070. PMID 32283783
- [Background] Palau-Rodriguez M, Garcia-Aloy M, Minarro A, Bernal-Lopez MR, Brunius C, Gomez-Huelgas R, Landberg R, Tinahones FJ, Andres-Lacueva C. Effects of a long-term lifestyle intervention on metabolically healthy women with obesity: Metabolite profiles according to weight loss response. Clin Nutr. 2020 Jan;39(1):215-224. doi: 10.1016/j.clnu.2019.01.018. Epub 2019 Feb 16. PMID 30862367
- [Background] Serrano JCE, Baena-Fustegueras JA, Martin-Gari M, Rassendren H, Cassanye A, Naudi A, Lopez-Cano C, Sanchez E, de la Fuente-Juarez MC, Herrerias Gonzalez F, Olsina Kissler JJ, Lecube A, Portero-Otin M. Adipose Tissue Protein Glycoxidation is Associated with Weight-Loss Potential. Obesity (Silver Spring). 2019 Jul;27(7):1133-1140. doi: 10.1002/oby.22501. Epub 2019 May 21. PMID 31112015
- [Background] Ciudin A, Fidilio E, Ortiz A, Pich S, Salas E, Mesa J, Hernandez C, Simo-Servat O, Lecube A, Simo R. Genetic Testing to Predict Weight Loss and Diabetes Remission and Long-Term Sustainability after Bariatric Surgery: A Pilot Study. J Clin Med. 2019 Jul 3;8(7):964. doi: 10.3390/jcm8070964. PMID 31277226
- [Background] Cornejo-Pareja I, Clemente-Postigo M, Tinahones FJ. Metabolic and Endocrine Consequences of Bariatric Surgery. Front Endocrinol (Lausanne). 2019 Sep 19;10:626. doi: 10.3389/fendo.2019.00626. eCollection 2019. PMID 31608009
- [Background] Arteaga-Gonzalez IJ, Martin-Malagon AI, Ruiz de Adana JC, de la Cruz Vigo F, Torres-Garcia AJ, Carrillo-Pallares AC. Bariatric Surgery Waiting Lists in Spain. Obes Surg. 2018 Dec;28(12):3992-3996. doi: 10.1007/s11695-018-3453-z. PMID 30121853
- [Background] Nicolau J, Simo R, Sanchis P, Ayala L, Fortuny R, Rivera R, Masmiquel L. Effects of depressive symptoms on clinical outcomes, inflammatory markers and quality of life after a significant weight loss in a bariatric surgery sample. Nutr Hosp. 2017 Feb 1;34(1):81-87. doi: 10.20960/nh.979. PMID 28244776
- [Background] Morcillo S, Martin-Nunez GM, Garcia-Serrano S, Gutierrez-Repiso C, Rodriguez-Pacheco F, Valdes S, Gonzalo M, Rojo-Martinez G, Moreno-Ruiz FJ, Rodriguez-Canete A, Tinahones F, Garcia-Fuentes E. Changes in SCD gene DNA methylation after bariatric surgery in morbidly obese patients are associated with free fatty acids. Sci Rep. 2017 Apr 10;7:46292. doi: 10.1038/srep46292. PMID 28393901